CLINICAL TRIAL: NCT01293565
Title: Evaluation of Phenotypic and Genetic Properties in Male Subjects Affected by Hypohidrotic Ectodermal Dysplasia
Brief Title: Evaluation of Phenotypic and Genetic Properties in Male Subjects Affected by Hypohidrotic Ectodermal Dysplasia - A
Status: Completed | Type: Observational
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ECP-003
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Hypohidrotic Ectodermal Dysplasia
Keywords: X-Linked Hypohidrotic Ectodermal Dysplasia; Hypohidrotic Ectodermal Dysplasia; XLHED; HED
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HED Affected Males
- Male Controls

SUMMARY:
The overall purpose of this study is to learn more about Hypohidrotic Ectodermal Dysplasia (HED) and to help in identifying treatment opportunities. Several evaluations will be conducted in this study: 1) the number of skin sweat glands you have and their ability to produce sweat; 2) your ability to grow hair; 3) the structure of your face compared to faces of people affected by HED; 4) molds of your teeth to see if and how they are different than people affected by HED.

ELIGIBILITY:
Inclusion Criteria:

1. Males age 14-29 years with clinical diagnosis of HED
2. No scalp shaving in the 6 months prior to enrollment
3. No current medical therapy for hair loss
4. Written informed consent for study and genotyping (or signed medical release of previous genetic test results)

Exclusion Criteria:

1. Medically significant condition as determined by the PI
2. Known hypersensitivity to pilocarpine or pilocarpine-like muscarinic agonists (e.g. Urecholine, Salagen, Pilocar, Provocholine)
3. Presence of cardiac pacemaker

Ages: 14 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: HED Affected Members of the UCSF Craniofacial Clinic, HED Affected Members of the National Foundation for Ectodermal Dysplasia
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To assess the hair follicle density and percent anagen hairs in the scalp of HED/XLHED males and unaffected controls | Day 1 and Day 3-4
To assess the palmar sweat duct number using confocal microscopy in HED/XLHED males and unaffected controls | Day 1
To evaluate 3-dimensional imaging technology without radiation exposure for mapping craniofacial development in HED/XLHED males and unaffected controls | Day 1
To use teeth impressions to construct 3-dimensional dental models for detailed evaluation of abnormalities present in HED/XLHED males (not for controls) | Day 1
To determine the presence or absence of EDA gene mutations/deletions in males with a clinical diagnosis of HED (not for controls) | Day 1
To assess by medical history the prevalence of medical complications in HED/XLHED males and unaffected controls | Day 1
To assess the pilocarpine-stimulated sweat rate on the volar surface of the forearm following pilocarpine iontophoresis in HED/XLHED males and unaffected controls, and to correlate with heat-stimulated sweat test classification | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Ophir Klein, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States